CLINICAL TRIAL: NCT02658552
Title: A Prospective Evaluation of High Intensity Focused Ultrasound (HIFU) in the Treatment of Benign Thyroid Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Lang Hung Hin, Brian, Clinical Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW15-486
Record Dates: First submitted 2016-01-06; First posted 2016-01-20 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Benign Thyroid Nodules
Keywords: HIFU; Benign thyroid nodule; Low risk; New treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HIFU treatment (Experimental): To collect the data after HIFU treatment
  Interventions: Device: Echopulse

INTERVENTIONS:
Device: Echopulse — Echopulse is a real-time US-guided High-intensity focused ultrasound (HIFU) system, the HIFU session is a noninvasive procedure that involves application of a focused high-energy ultrasound beam for thermal tissue ablation inside the targeted zone, with minimal effect on the surrounding tissue

SUMMARY:
To evaluate the short-term efficacy of high intensity focused ultrasound (HIFU) in the treatment of benign thyroid nodules

DETAILED DESCRIPTION:
Background:

Thyroid nodules are very common worldwide. In an iodine-replete population like Hong Kong, the estimated prevalence of a clinically palpable thyroid nodule, is close to 5% while the prevalence of ultrasonically detectable nodules could be up to 67%. With the frequent use of computed tomography, carotid ultrasound studies and positron emission scans nowadays, many small, non-palpable thyroid nodules are incidentally detected. The use of high intensity focused ultrasound MRI guided or ultrasound guided have been used to treat different types of soft tissue cancer like prostate cancer, liver cancer and breast cancer. This device has been tried in a clinical study where patients with thyroid nodules, who were already scheduled for thyroidectomy, were treated using HIFU in order to evaluate the safety and feasibility of the device and to better determine the treatment parameters and effect.

The results showed that the overall safety of the treatment was satisfactory and the lesions produced by the HIFU shots in the nodule were precise. This pilot study was extended to a clinical trial where patients with a benign thyroid nodule were treated. Twenty-one patients were treated in this study versus 11 controls. No serious adverse events (SAE) have occurred. A patient with a toxic thyroid nodule was also treated with the HIFU device (Theraclion, France). The treatment was well tolerated and biologic euthyroidism was achieved at 3 months (TSH, 1.91 mIU/L) and was maintained at 6, 12, and 18 months. At 12 and 18 months, the treated nodule was barely seen as a nonvascularized hypoechoic scar. Thyroid scintigraphy showed a recovery of the thyroid iodine uptake.

Since November 1st 2007, this HIFU device (Theraclion, France) has been CE marked for HIFU treatment of neck pathologies. 11 patients with primary hyperparathyroidism have been treated and followed. The mean follow-up is 9.5 months (1-28 months).

Symptomatic hypocalcaemia was not observed in any patient after HIFU treatments or during follow-up. A prospective monocenter study was performed in Bulgaria for the treatment of benign solid thyroid nodule by US-Guided HIFU. Twenty thyroid nodules were treated during one HIFU session. The mean ± standard deviation nodule volume was 4.96 mL ± 2.79 at the start of the study. Nodule volume had decreased to 3.05 mL ±1.96 at the 3-month follow-up examination (n = 20, P < .001), and reached 2.91 mL ± 2.43 by the 6-month follow-up examination (n = 16, P < .001). By then, the mean volume reduction was 48.7% ± 24.3 (P< .001). Minor transient complications such as subcutaneous edema and mild skin redness were observed in two patients. Another monocenter study was performed in Germany in 2014. Ten patients with one thyroid nodule each were treated by HIFU. Three months after the procedure, thyroid nodule volume was significantly reduced by 48.8% (median) and a shrinkage up to 75% of the volume was observed. In terms of safety, no serious side effect related to the procedure was reported.

Objectives:

The present study is aimed to explore the followings:

1. To evaluate the efficacy of the HIFU for the treatment of benign thyroid nodules using assessment of patient experience and adverse event reporting.
2. To evaluate the tolerance of HIFU in the treatment of benign thyroid nodules.
3. To determine the location parameters associated with optimal efficiency tissue ablation.

The procedure schedule comprises:

* An first visit (V0)
* The HIFU session (D0)
* A visit at 1, 3 and 7 days after HIFU session (D1, D3, D7)
* A visit at 3 and 6 months (M3, M6).
* At each visit: any local and/or general adverse event will be documented in case report form (CRF).

Ultrasound measurement of the treated nodule (in 3 dimensions) will be performed at each scheduled visit.

The treatment procedure of Echopulse consists of five treatment steps:

* Pre-treatment ultrasonography
* Positioning
* Planning
* Generation of HIFU treatment pulses in the volume defined above; power setting is achieved on regularly spaced sites subsets.
* Post-treatment visualization and final report. The parameters of HIFU treatment will be part of the clinical study data base. When an HIFU session is prematurely interrupted, the reason of interruption will be recorded in the CRF (adverse event, technical failure, others).

Study duration will lbe 6 months for each patient, counting from the post-HIFU day.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient 18 years or older.
* Patient presenting with at least one thyroid nodule with no signs of malignancy:

  1. Non suspicious clinically and at ultrasonography imaging
  2. Benign cytological diagnosis at fine needle aspiration biopsy in the last 6 months
  3. Normal serum calcitonin
  4. No history of neck irradiation
* Serum TSH and free T4 levels within the normal range
* Targeted nodule deemed to be accessible and eligible to HIFU
* Absence of vocal cord paresis at laryngoscopy
* Nodule greatest diameter between ≥10 - 20mm as measured by ultrasound
* Composition of the targeted nodule(s) : predominantly solid
* Patient is mentally competent and has given informed consent.

Exclusion Criteria:

* Head and/or neck disease that prevents extension of neck
* Known history of thyroid cancer or other malignant tumors in the neck region
* History of neck irradiation
* Intranodular macrocalcification inducing a shadow in the thyroid significant enough to preclude HIFU treatment
* A nodule next to the posterior margin of the lobe with distance <15mm
* Pregnant or lactating woman
* Any contraindication to the assigned analgesia/anaesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-10; Primary Completion 2016-02 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The changing volume of benign thyroid nodule after HIFU treatment | 6 months
  Change in volume (ml) of the targeted benign thyroid nodule 6 months after one successful course of HIFU
The changing greatest dimension of benign thyroid nodule after HIFU treatment | 6 months
  Change in greatest dimension (in mm) of the targeted benign thyroid nodule 6 months after one successful course of HIFU

SECONDARY OUTCOMES:
The pain assessment (scoring 1-10) after treatment | 6 months
  Patient pain score immediately after completion of HIFU treatment session.
Incidence of local/ or general adverse events | 6 months
  The incidence rate of local or general adverse events after completion of HIFU treatment session.

CONTACTS AND LOCATIONS:
Overall Officials: Hung Hin, Brian Lang, MBBS(Hons), Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Hegedus L, Bonnema SJ, Bennedbaek FN. Management of simple nodular goiter: current status and future perspectives. Endocr Rev. 2003 Feb;24(1):102-32. doi: 10.1210/er.2002-0016. PMID 12588812
- [Background] Erdogan MF, Gursoy A, Erdogan G. Natural course of benign thyroid nodules in a moderately iodine-deficient area. Clin Endocrinol (Oxf). 2006 Dec;65(6):767-71. doi: 10.1111/j.1365-2265.2006.02664.x. PMID 17121528
- [Background] Bergenfelz A, Jansson S, Kristoffersson A, Martensson H, Reihner E, Wallin G, Lausen I. Complications to thyroid surgery: results as reported in a database from a multicenter audit comprising 3,660 patients. Langenbecks Arch Surg. 2008 Sep;393(5):667-73. doi: 10.1007/s00423-008-0366-7. Epub 2008 Jul 17. PMID 18633639
- [Background] Sung JY, Baek JH, Kim KS, Lee D, Yoo H, Kim JK, Park SH. Single-session treatment of benign cystic thyroid nodules with ethanol versus radiofrequency ablation: a prospective randomized study. Radiology. 2013 Oct;269(1):293-300. doi: 10.1148/radiol.13122134. Epub 2013 Apr 24. PMID 23616630
- [Background] Gharib H, Hegedus L, Pacella CM, Baek JH, Papini E. Clinical review: Nonsurgical, image-guided, minimally invasive therapy for thyroid nodules. J Clin Endocrinol Metab. 2013 Oct;98(10):3949-57. doi: 10.1210/jc.2013-1806. Epub 2013 Aug 16. PMID 23956350
- [Background] Baek JH, Lee JH, Valcavi R, Pacella CM, Rhim H, Na DG. Thermal ablation for benign thyroid nodules: radiofrequency and laser. Korean J Radiol. 2011 Sep-Oct;12(5):525-40. doi: 10.3348/kjr.2011.12.5.525. Epub 2011 Aug 24. PMID 21927553
- [Background] Zhou YF. High intensity focused ultrasound in clinical tumor ablation. World J Clin Oncol. 2011 Jan 10;2(1):8-27. doi: 10.5306/wjco.v2.i1.8. PMID 21603311
- [Background] Kovatcheva RD, Vlahov JD, Shinkov AD, Borissova AM, Hwang JH, Arnaud F, Hegedus L. High-intensity focused ultrasound to treat primary hyperparathyroidism: a feasibility study in four patients. AJR Am J Roentgenol. 2010 Oct;195(4):830-5. doi: 10.2214/AJR.09.3932. PMID 20858805
- [Background] Kovatcheva RD, Vlahov JD, Stoinov JI, Kirilov GG, Krivoshiev SG, Arnaud F, Ortuno C, Drueke TB. High-intensity focussed ultrasound (HIFU) treatment in uraemic secondary hyperparathyroidism. Nephrol Dial Transplant. 2012 Jan;27(1):76-80. doi: 10.1093/ndt/gfr590. Epub 2011 Oct 19. PMID 22015443
- [Background] Kovatcheva R, Vlahov J, Stoinov J, Lacoste F, Ortuno C, Zaletel K. US-guided high-intensity focused ultrasound as a promising non-invasive method for treatment of primary hyperparathyroidism. Eur Radiol. 2014 Sep;24(9):2052-8. doi: 10.1007/s00330-014-3252-4. Epub 2014 Jun 4. PMID 24895038
- [Background] Esnault O, Franc B, Monteil JP, Chapelon JY. High-intensity focused ultrasound for localized thyroid-tissue ablation: preliminary experimental animal study. Thyroid. 2004 Dec;14(12):1072-6. doi: 10.1089/thy.2004.14.1072. PMID 15650361
- [Background] Esnault O, Franc B, Chapelon JY. Localized ablation of thyroid tissue by high-intensity focused ultrasound: improvement of noninvasive tissue necrosis methods. Thyroid. 2009 Oct;19(10):1085-91. doi: 10.1089/thy.2009.0121. PMID 19803790
- [Background] Esnault O, Franc B, Menegaux F, Rouxel A, De Kerviler E, Bourrier P, Lacoste F, Chapelon JY, Leenhardt L. High-intensity focused ultrasound ablation of thyroid nodules: first human feasibility study. Thyroid. 2011 Sep;21(9):965-73. doi: 10.1089/thy.2011.0141. Epub 2011 Aug 11. PMID 21834683
- [Background] Esnault O, Rouxel A, Le Nestour E, Gheron G, Leenhardt L. Minimally invasive ablation of a toxic thyroid nodule by high-intensity focused ultrasound. AJNR Am J Neuroradiol. 2010 Nov;31(10):1967-8. doi: 10.3174/ajnr.A1979. Epub 2010 Jan 14. PMID 20075098
- [Background] Huh JY, Baek JH, Choi H, Kim JK, Lee JH. Symptomatic benign thyroid nodules: efficacy of additional radiofrequency ablation treatment session--prospective randomized study. Radiology. 2012 Jun;263(3):909-16. doi: 10.1148/radiol.12111300. Epub 2012 Mar 21. PMID 22438360
- [Background] Vitti P, Rago T, Mazzeo S, Brogioni S, Lampis M, De Liperi A, Bartolozzi C, Pinchera A, Martino E. Thyroid blood flow evaluation by color-flow Doppler sonography distinguishes Graves' disease from Hashimoto's thyroiditis. J Endocrinol Invest. 1995 Dec;18(11):857-61. doi: 10.1007/BF03349833. PMID 8778158